CLINICAL TRIAL: NCT01574027
Title: Efficacy of Vitamin D in Colorectal Cancer Chemoprevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Richard Benya, M.D., MD, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01CA122299 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Colorectal Cancer
Keywords: Assess the efficacy of vitamin D for preventing colorectal cancer and identifying the populations likely (or unlikely) to benefit from vitamin D-based therapy.; Evaluate the ability of Vitamin D3 (cholecalciferol) to reduce ACF's in humans.
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Some participants were given a placebo pill to take daily for the length of the study. The placebo patients were used as a control group to compare against those taking the Vitamin D supplement.
  Interventions: Drug: Placebo
- Vitamin D3 (cholecalciferol) (Experimental): Other participants were administered Vitamin D3 (cholecalciferol) for the six month study duration to determine if it would decrease the number of aberrant crypt foci in the colon as compared to the baseline number.
  Interventions: Drug: Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Drug: Vitamin D3 (cholecalciferol) — One capsule per day for six months
  Arms: Vitamin D3 (cholecalciferol)
Drug: Placebo — One capsule per day for six months
  Arms: Placebo

SUMMARY:
Vitamin D's ability to prevent colorectal cancer (CRC) has been suspected for nearly 30 years, but has never been directly studied in humans. The biologically active version of vitamin D, 1,25(OH)2D3, cannot be readily used in humans because of its tendency to cause serum calcium levels to rise. In contrast, 25(OH)D3 (ie calcifediol) does not have this side effect. The investigators previous research suggests that the enzyme necessary to convert 25(OH)D3 (calcifediol) into active 1,25(OH)D3 is present in cells lining the large intestine (colon).

Aberrant crypt foci (ACF) are very small (ie microscopic) collections of abnormally shaped cells that are a commonly used marker of CRC risk. Screening colonoscopy at UIC routinely uses methods that allow ACF counting to be done as a part of standard practice. ACF's are not fixed, like polyps or cancers, but can disappear as a person's risk for developing CRC decreases.

The investigators propose giving patient's with 10 or more ACF's 25(OH)D3 (calcifediol) or placebo, and determining if there is a drug-dependant decrease in ACF number. The primary objective is to determine whether 25(OH)D3 (calcifediol) supplementation, compared to placebo, causes significant reduction of ACF number from baseline levels. The primary endpoint will be change in ACF number.

DETAILED DESCRIPTION:
Patients will be offered participation in this study at the time of their regularly scheduled visit to the UIC Colorectal Cancer Screening Clinic. Those agreeing will have indicated their understanding that participation will be conditional upon their having 10+ ACF at the time of their screening colonoscopy. If at screening colonoscopy 10+ ACF are found patients will:

* undergo 3 endoscopic mucosal biopsies of the distal colon; and
* undergo a blood draw from an i.v. already in place for sedative-narcotic administration for serum 25(OH)D3 and serum ionized calcium; and
* be given either placebo or calcifediol and instructed to take daily for 6 months.
* provide urine for calcium/creatine spot ratio.

At 7 and 14 days after the screening colonoscopy patients will be called on the telephone by the clinical research nurse assigned to this study to follow-up and note 25(OH)D3 (calcifediol) toxicity, if any (note that toxicity has not been described except in the case of overdose). Signs specifically looked for will include: headache, increased urination, nausea, vomiting, abdominal pain, weakness, constipation, and anorexia. If present, patient will be advised to present immediately to the UIC GCRC for physical and serological evaluation.

At 30, 90 and 120 days the patient will have agreed to present to the GCRC clinic for:

* Capsule retrieval/count (80% compliance will be required to remain in study); and
* Detailed history and physical, focusing specifically on signs and symptoms of hypercalcemia.
* At day 90 only - provide urine for calcium/creatine spot ratio.

Evidence on exam, or laboratory, of hypercalcemia will result in an adverse event reporting and immediate patient discharge from this study. Signs specifically looked for include: headache, increased urination, nausea, vomiting, abdominal pain, weakness, constipation, and anorexia.

At 180 days the patient will have agreed to undergo:

* Repeat endoscopic exam limited to the recto-sigmoid colon, also known as a "flexible sigmoidoscopy"; and
* repeat blood draw for serum 25(OH)D3 and serum ionized calcium

ELIGIBILITY:
Inclusion Criteria:

* All non-pregnant patients 50 years of age or older with 10 or more ACFs.

Exclusion Criteria:

* The following will be specifically looked for, and result in patients not being eligible for study enrollment:
* Use of non-steroidal anti-inflammatory drugs or glucocorticosteroids within 60 days of study entry.
* History of chronic IBD or prior pelvic radiation (inflammation distorts crypt pattern).
* Intake of any vitamin D or calcium supplements within 60 days of study entry.
* Patients with increased bleeding risk from biopsy protocol (i.e. renal failure, decompensated cirrhosis, blood dyscrasia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Reduction in ACF biomarkers | 6 months
  The investigators propose giving patient's with 10 or more ACF's 25(OH)D3 (calcifediol) or placebo, and determining if there is a drug-dependant decrease in ACF number. The primary objective is to determine whether 25(OH)D3 (calcifediol) supplementation, compared to placebo, causes significant reduction of ACF number from baseline levels. The primary endpoint will be change in ACF number.

CONTACTS AND LOCATIONS:
Overall Officials: Richard V Benya, M.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Medical Center, Chicago, Illinois, United States